CLINICAL TRIAL: NCT04749420
Title: Translation, Cultural Adaptation, Reliability, and Validity of the Turkish Version of the Cervical Radiculopathy Impact Scale
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ARIKAN, Research Assistant, Gazi University
Other Study IDs: 26.01.2021-E.13997
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Cervical Radiculopathy; Cervical Radicular Pain; Cervical Radiculitis; Cervical Root Syndrome
Keywords: Cervical radiculopathy; Reliability; Validity; Cross-cultural adaptation
MeSH Terms: conditions — Radiculopathy | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients group: Individuals with cervical radiculopathy
  Interventions: Other: Survey study

INTERVENTIONS:
Other: Survey study — Cervical Radiculopathy Impact Scale (CRIS) will be applied

SUMMARY:
The purpose of this study was to investigate adaptation, validity, and reliability of the Turkish version of the Cervical Radiculopathy Impact Scale (CRIS).

DETAILED DESCRIPTION:
Cervical radicular syndrome is a common health problem that causes pain in the arm and / or hand and is accompanied by motor and / or sensory defects. These symptoms often have an intensity that prevents normal function. For individuals with cervical radicular syndrome, there is a lack of a patient-reported outcome measurement tool to measure the impact of the disorder. The Cervical Radiculopathy Impact Scale (CRIS), which focuses on the symptoms and functionality of the arm and neck, was developed to improve the quality of studies on cervical radicular syndrome. CRIS is a newly developed self-report questionnaire that covers the measurement of symptoms and limitations in individuals with cervical radiculopathy due to pain, tingling sensation, and loss of sensation in the arm with neck discomfort. The CRIS consists of 21 items divided into three subscales: (i) symptoms, (ii) energy and postures, and (iii) actions and activities. Each item contains a likert type answer and takes a value between 1 and 5. The study is planned with 105 individuals with hip disease. After questioning the sociodemographic characteristics of the individuals, the patients will be asked to fill in CRIS, EQ-5D Health-Related Quality of Life Questionnaire, Neck Disability Index, Quick Disabilities of the Arm Shoulder and Hand, Brief Illness Perception Questionnaire, Short Form-36 and Visual Analog Scale. Test-retest will be re-applied to those of the same individuals who can be reached after 1 week. The results will be analyzed using the SPSS version 22.0 computer package program.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with radiculopathy symptoms and diagnosis.

Exclusion Criteria:

* Having another neck disorder other than radiculopathy,
* History of cervical spine surgery,
* Corticosteroid injection to cervical spine in the past 3 months,
* Having neurological and cognitive disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals with cervical radiculpathy symptoms, diagnosis, and chronic pain on cervical spine region.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Cervical Radiculopathy Impact Scale (CRIS) | 12 minutes
  Cervical Radiculopathy Impact Scale was designed to evaluate measurement of symptoms and limitations in individuals with cervical radiculopathy.

CONTACTS AND LOCATIONS:
Locations (1):
- Halime ARIKAN, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR